CLINICAL TRIAL: NCT01551862
Title: Prospective Study on Complications Following a Lower Body Lift After Massive Weight Loss
Brief Title: Complications in Lower Body Lifts
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Hugo B. Kitzinger, Principal investigator, Medical University of Vienna
Other Study IDs: PlastSurg01
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Surplus Skin After Massive Weight Loss
Keywords: lower body lift; body contouring surgery; massive weight loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: body contouring surgery of back, abdomen and thighs — simultaneous body contouring surgery of back, abdomen and thighs

SUMMARY:
A prospective study on 50 consecutive patients who are going to have a lower body lift procedure is performed. Measures include comorbidities and complications. Risk factors assessed including patient age, gender, highest lifetime body mass index (BMI) (BMI max), current BMI, excess weight loss (EWL), type of weight loss and nicotine consumption.

ELIGIBILITY:
Inclusion Criteria:

* after massive weight loss
* age > 18 years and < 65 years
* excess weight loss > 66%
* current body mass index < 35
* stable weight after weight loss for at least 12 months

Exclusion Criteria:

* insulin dependent diabetes mellitus

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients which are referred to Department of Plastic Surgery for body contouring surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo B Kitzinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dept. of Plastic Surgery, Vienna, Austria

REFERENCES:
- [Derived] Kitzinger HB, Cakl T, Wenger R, Hacker S, Aszmann OC, Karle B. Prospective study on complications following a lower body lift after massive weight loss. J Plast Reconstr Aesthet Surg. 2013 Feb;66(2):231-8. doi: 10.1016/j.bjps.2012.09.006. Epub 2012 Oct 4. PMID 23040202